CLINICAL TRIAL: NCT05854654
Title: Defining Novel Strategies for the Diagnosis and Treatment of Intraoperative Air Leaks: An Ex-Vivo Human Lung Model Study
Brief Title: Air Leak Detection and Treatment
Acronym: CT0128
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-11357
Record Dates: First submitted 2023-04-13; First posted 2023-05-11 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Air Leak From Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air Leaks (Experimental): Lungs from patients undergoing lung transplantation after their removal from the recipient patient with previous informed consent signed before transplantation will be obtained. The organs will be placed in an acrylic box and will be kept at a temperature of 37 Celsius degrees. In order to reproduce intraoperative air leaks, various manipulations, including stapling and creating lacerations of different depts and lengths on the parenchyma, will be performed on deflated lungs. Following the introduction of a leak, condensed gas will be pushed through the airway to precisely localize the defect. The sealant prepared at room temperature will then be applied in a thin layer to cover the defect and will be left to dry for 5 minutes. The seal will be tested using the condensed gas with the lung still deflated as well as with the water immersion technique after inflating the lung.
  Interventions: Diagnostic Test: Air Leaks

INTERVENTIONS:
Diagnostic Test: Air Leaks — The organs will be placed in an acrylic box and will be kept at a temperature of 37 Celsius degrees. The lungs will be mechanically ventilated connected by an endotracheal tube size 8 inserted in the bronchus with the balloon inflated and a silk suture providing an hermetic closure proximal to the balloon.
  This setting will allow us to perform several different endoscopic and RAB procedures in emulated physiologic conditions to complete the study.

SUMMARY:
Developing a methodology to detect, quantify and treat air leaks intraoperatively using a bio-adhesive, to thereby reduce postoperative surgical complications, morbidity, and length of stay for patients undergoing pulmonary resection.

DETAILED DESCRIPTION:
This study aims at establishing a standardized, stable and effective ex-vivo human lung model, applying some changes to settings used in our previous studies both in animal and human models performed in this institution. Multiple procedures will be performed to each model in order to accomplish the objectives of the study. Tissue samples will be taken from the models and images will be performed. This will allow us to determine which configuration is the optimal for obtaining the more effective and stable models that could offer the best quality specimens as well. Lungs from patients undergoing lung transplantation after their removal from the recipient patient with previous informed consent signed before transplantation will be obtained. The organs will be placed in an acrylic box and will be kept at a temperature of 37 Celsius degrees. The lungs will be mechanically ventilated connected by an endotracheal tube size 8 inserted in the bronchus with the balloon inflated and a silk suture providing an hermetic closure proximal to the balloon. Alternatively, and as performed in one of our previous studies, according to the bronchial stump length and diameter, a Penrose drain (1 inch) will be sewn to the mainstem bronchus to simulate the trachea and allow for an endotracheal tube (ET), size 9.0 Fr, to be inserted into and secured with the Penrose drain. Following, a Sheridan® Sher-I-SWIV/FO ™ Double Swivel Connector will be inserted to the tube to allow performing endoscopic and RAB procedures while maintaining ventilation. The mechanical ventilator will be set using positive pressure and high tidal volume to prevent the lungs from collapsing.

A cannula will be placed in the pulmonary artery and secured with a purse-string suture. The lung will be perfused with 37°C solution using a roller pump (Terumo Sarns, Tokyo, Japan) with a flow rate (usually ~0.2 L/min) was adjusted to maintain a pulmonary arterial pressure of 10-12 mmHg to prevent hydrostatic pulmonary edema. The pulmonary veins will not be cannulated, allowing the perfusate to drain passively from the pulmonary veins into the reservoir at the base of the acrylic chamber from where it will be recycled through the pump. Temperatures of the lung tissue, ambient, container, and intravascular will be monitored by thermocouples. The pulmonary arterial pressure will be measured via a pulmonary arterial catheter (Cook, Bloomington, IN) placed in the circuit at the level of the left atrium. Once the model reaches a stable temperature 36°C, the procedures will begin.

This setting will allow us to perform several different endoscopic and RAB procedures in emulated physiologic conditions to complete the study.

In order to reproduce intraoperative air leaks, various manipulations, including stapling and creating lacerations of different depts and lengths on the parenchyma, will be performed on deflated lungs. Following the introduction of a leak, condensed gas will be pushed through the airway to precisely localize the defect. The sealant prepared at room temperature will then be applied in a thin layer to cover the defect and will be left to dry for 5 minutes. The seal will be tested using the condensed gas with the lung still deflated as well as with the water immersion technique after inflating the lung.

The leaks will be quantified using the Thopaz automated drainage system by Medela.

In order to test the long term stability of the matrix, the lung will be ventilated for X minutes. Air leak testing will be repeated at specific intervals during this time.

After all the procedures are finished and specimens obtained, all the lungs will be sent to the CHUM and will be processed following the standard hospital protocol for transplants recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lung transplant surgery
* Organ donor ineligible to donate lungs

Exclusion Criteria:

* Healthy individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Detection and localisation of air leaks in deflated lungs using condensed air through the airway. Changing the size (ml) of air leaks by 80% by the use of a novel bio sealant directly on the lung parenchyma. | 48 months
  The evaluation of different techniques for the detection and localisation of air leaks in deflated lungs.
  The application of the novel bio sealant on staple lines or localized lacerations on the lung parenchyma from instrumentation or other will result in a change in the volume (ml) of air leaks.

SECONDARY OUTCOMES:
Establishing a standardized measure to localize air leaks in a physiological setting. | 48 months
  Based on preliminary findings, a standardized methodology for the localization will be established
Quantify and treat air leaks in a physiological setting | 48 months
  Time to seal air leaks Quantity of air leaks Seal percentage change in output of leak (measured in mL/min)
Quantify and treat air leaks in a physiological setting | 48 months
  Comparison in effectiveness of varying sealing technologies Optimal methods for application of sealant Sealant loss (% of total applied)

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, Principal Investigator — CHUM
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No